CLINICAL TRIAL: NCT00244335
Title: Emotional Control of Sedative Self-Medication in Post-Traumatic Stress Disorder
Brief Title: Examining the Role of Negative Emotional States on Sedative Drug Use in Individuals With Post-Traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: John Casada, MD, PhD/Pedro Delgado, MD, Chairman, University of Texas Health Science Center at San Antonio
Other Study IDs: NIDA-00507-1; K08-00507-1; DPMC
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-08

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post-Traumatic Stress Disorders; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: PTSD Subjects
- 2: Trauma Controls: subjects who have experienced a trauma but never developed PTSD

SUMMARY:
Post-traumatic stress disorder (PTSD) is a serious illness, in which individuals often experience anxiety and stress. Some individuals with PTSD use drugs to alleviate emotional distress. This study will examine the role that negative emotional states play in sedative drug use among individuals with PTSD.

DETAILED DESCRIPTION:
PTSD is a psychiatric illness that occurs following a traumatic event in which there was threat of injury or death to an individual. Common symptoms of PTSD include anxiety, stress, and tension. Some individuals with PTSD use benzodiazepines, a type of sedative medication, or alcohol to alleviate the anxiety associated with the disorder. Past research has shown that the negative feelings experienced by individuals with PTSD may increase the reinforcing effects of antidepressant drugs. Feelings of anxiety act as a stimulus, which leads to drug use; in turn, the anticipated or actual decrease in distress reinforces the drug-taking behavior. Greater amounts of sedative drugs are then needed to decrease subsequent stress and anxiety. The purpose of this study is to understand how negative emotional states affect the reinforcing effects of sedative drugs in individuals with PTSD.

This study will enroll two types of individuals, both of whom have been exposed to an emotional trauma and report using alcohol to reduce emotional distress but who differ in their subsequent development of PTSD. Participants will take part in an initial screening session which will include a physical examination, standardized psychological questionnaires, and review of medical and drug histories. Once enrolled, each participant will take part in 8 experimental session days, with each day of testing separated by at least 48 hours. At the beginning of each session, a breathalyzer and urine test will be used to screen for the presence of alcohol and drugs. On Day 1, participants will take part in an orientation session to familiarize themselves with the laboratory and study procedures. On Days 2 through 4, participants will receive varying doses of alcohol, a placebo drink, a placebo drug, and alprazolam, a type of benzodiazepine medication. On Days 5 through 8, participants will take part in experimental challenges designed to induce various emotional states, including arousal, anxiety, aggression, and anger. They will also complete a monetary reward task to measure the reinforcing effects of drugs. Participants will complete questionnaires several times each day to assess anxiety, anger, drug effects, and drug cravings. Heart rate will be monitored with an electrocardiogram, and electrodes placed on the skin will measure other physiologic measures throughout each session. Participants will receive compensation for completing each experimental session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD with anxiety symptoms, as determined by a score greater than 14 on the Hamilton Anxiety Rating Scale, or a score greater than 18 on the Profile of Mood States-Tension Anxiety Rating Scale
* Experiences frequent and intense PTSD symptoms
* Able to spend 6 hours at a time in the research laboratory
* If a trauma control participant, must have experienced a trauma that meets criterion A for PTSD, but has never developed PTSD
* Willing to use contraception throughout the study

Exclusion Criteria:

* Females who meet DSM-IV diagnostic criteria for premenstrual dysphoric disorder
* Females who report premenstrual distress that motivates them to use alcohol for relief
* History of bipolar affective disorder, any psychotic disorder, current major depressive episode, or current primary non-PTSD anxiety disorder (individuals with Axis II diagnoses will not be excluded)
* Currently enrolled in psychodynamic or cognitive-behavioral therapy
* Current unstable medical illness
* Current medical illness treated with psychoactive drugs (e.g., beta blockers)
* Current medical illness with complicating psychiatric symptoms (e.g., thyroid disease)
* Requires use of certain medications
* Current or past history of illicit substance dependence, other than past marijuana abuse or dependence
* History of tobacco dependence
* Failure to provide a drug-free urine sample prior to study entry
* Smokes more than one pack of cigarettes per day or drinks beverages totaling more than 500 mg of caffeine per day
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: PTSD subjects and subjects who have experienced a trauma but never developed PTSD (Trauma Controls) are being recruited for this study. Recruitment is being conducted through Audie L. Murphy Veterans Administration Hospital and the University of Texas Health Science Center at San Antonio.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2000-10; Primary Completion 2006-02 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Casada, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Result] Casada JH, Roache JD. Dissociation of physiology and behavior in PTSD. Int J Psychophysiol. 2006 Nov;62(2):243-8. doi: 10.1016/j.ijpsycho.2006.04.005. Epub 2006 Jul 11. PMID 16814888
- [Result] Casada JH, Roache JD. Behavioral inhibition and activation in posttraumatic stress disorder. J Nerv Ment Dis. 2005 Feb;193(2):102-9. doi: 10.1097/01.nmd.0000152809.20938.37. PMID 15684912